CLINICAL TRIAL: NCT00879814
Title: A Phase 1 Randomized, Open-label, Parallel-group, Active- And Placebo-controlled Study To Assess Safety And Tolerability Of 60, 120, And 200 Mcg Meningococcal Group B Rlp2086 Vaccine In Healthy Adult Subjects
Brief Title: Study Evaluating Safety And Tolerability Of Meningococcal B Rlp2086 Vaccine In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6108A1-1004; B1971004 (Other: Alias Study Number)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-07

CONDITIONS: Meningitis, Meningococcal
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): rLP2086 vaccine 60 mcg
  Interventions: Biological: rLP2086 vaccine or control
- 2 (Experimental): rLP2086 vaccine 120 mcg
  Interventions: Biological: rLP2086 vaccine or control
- 3 (Experimental): rLP2086 vaccine 200 mcg
  Interventions: Biological: rLP2086 vaccine or control
- 4 (Active Comparator): Tdap vaccine - normal saline - normal saline
  Interventions: Biological: rLP2086 vaccine or control

INTERVENTIONS:
Biological: rLP2086 vaccine or control — intra-muscular vaccine (solution), 0.5 mL, 3 doses, schedule: 0, 2, 6 months
  Arms: 1
Biological: rLP2086 vaccine or control — intra-muscular vaccine (solution), 0.5 mL, 3 doses, schedule: 0, 2, 6 months
  Arms: 2
Biological: rLP2086 vaccine or control — intra-muscular vaccine (solution), 0.5 mL, 3 doses, schedule: 0, 2, 6 months
  Arms: 3
Biological: rLP2086 vaccine or control — intra-muscular vaccine (solution), 0.5 mL, 3 doses, schedule: 0, 2, 6 months
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of an investigational meningococcal B rLP2086 vaccine in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet the following inclusion criteria at screening (visit 1) and at randomization (visit 2) to be considered for enrollment in the study:

* Male or female subjects between the ages of 18 and 40.
* Healthy male or female subjects as determined by medical history, physical examination, and judgment of the investigator.
* Male or female subject who is considered biologically capable of having children must agree to commit to the use of a reliable method of birth control for the duration of the study and for 30 days after early discontinuation. A subject is still biologically capable of having children, even if he or she is using contraceptives or if his or her sexual partner is sterile or using contraceptives.

In addition a subject must meet the following inclusion criteria at randomization (visit 2) to be considered for enrollment in the study. The referred blood and urinalysis tests (inclusion criterion 5) will be performed on a blood and urine sample taken at visit 1:

* Female subjects of childbearing potential with a negative urine pregnancy test prior to study drug administration. Note: this criterion will apply to each vaccination visit and to the last study visit.
* Laboratory blood and urinalysis tests results within the per-protocol normal ranges.
* Able to be contacted by telephone during the study period. Note: this criterion will apply to each study visit.

Exclusion Criteria:

None

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Miami Research Associates, Inc., South Miami, Florida, United States

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Sheldon EA, Schwartz H, Jiang Q, Giardina PC, Perez JL. A phase 1, randomized, open-label, active-controlled trial to assess the safety of a meningococcal serogroup B bivalent rLP2086 vaccine in healthy adults. Hum Vaccin Immunother. 2012 Jul;8(7):888-95. doi: 10.4161/hv.19983. Epub 2012 Jul 1. PMID 22832260
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6108A1-1004&StudyName=Study%20Evaluating%20Safety%20And%20Tolerability%20Of%20Meningococcal%20B%20Rlp2086%20Vaccine%20In%20Healthy%20Adults

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 189 participants who signed informed consent form, 134 were screen failures (mainly because of laboratory abnormalities) and 7 participants withdrew before the first vaccination. Total 48 participants were randomized into 4 groups.
Groups:
- rLP2086 60mcg; rLP2086 120 mcg; rLP2086 200 mcg: Given on a 0, 2-, 6- month schedule
- Tdap/Normal Saline (Control): Tdap was given at month 0 and Saline was given at Month 2 and 6
Period: Overall Study
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Started | 12 | 12 | 12 | 12
Completed | 8 | 10 | 9 | 7
Not Completed | 4 | 2 | 3 | 5
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2
Not completed — Participant Failed to Return | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (7.40) | 31.0 (7.65) | 27.8 (6.05) | 27.2 (5.77) | 28.8 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 10 | 7 | 29
  Male | 6 | 6 | 2 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants | 91.7 | 91.7 | 91.7 | 91.7

2. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Alanine Aminotransferase [ALT])
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 91.7 | 83.3 | 91.7
  Baseline: Normal, Post-Baseline: Mild | 0 | 8.3 | 16.7 | 8.3

3. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Aspartate Aminotransferase [AST])
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 91.7 | 100.0 | 91.7
  Baseline: Normal, Post-Baseline: Mild | 0 | 8.3 | 0 | 0
  Baseline: Normal, Post-Baseline: Moderate | 0 | 0 | 0 | 8.3

4. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Total Protein)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 100.0 | 100.0
  Baseline:Normal,Post Baseline:Mild/Moderate/Severe | 0.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Albumin)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 100.0 | 100.0
  Baseline:Normal,Post Baseline:Mild/Moderate/Severe | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Alkaline Phosphatase [ALP])
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 91.7 | 100.0 | 100.0
  Baseline: Normal, Post-Baseline: Mild | 0 | 8.3 | 0 | 0

7. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Total Bilirubin)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 91.7 | 100.0 | 91.7
  Baseline: Normal, Post-Baseline: Moderate | 0 | 8.3 | 0 | 0
  Baseline: Normal, Post-Baseline: Grade 4 | 0 | 0 | 0 | 8.3

8. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Creatine Phosphokinase [CPK])
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 91.7 | 91.7 | 75.0
  Baseline: Normal, Post-Baseline: Mild | 0 | 0 | 8.3 | 0
  Baseline: Normal, Post-Baseline: Moderate | 0 | 8.3 | 0 | 16.7
  Baseline: Normal, Post-Baseline: Grade 4 | 0 | 0 | 0 | 8.3

9. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Prothrombin Time [PT])
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 91.7 | 100.0
  Baseline: Normal, Post-Baseline: Moderate | 0 | 0 | 8.3 | 0

10. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Partial Thromboplastin Time [PTT])
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 83.3 | 50.0 | 50.0 | 75.0
  Baseline: Normal, Post-Baseline: Mild | 16.7 | 50.0 | 33.3 | 25.0
  Baseline: Normal, Post-Baseline: Moderate | 0 | 0 | 16.7 | 0

11. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Fibrinogen)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 83.3 | 75.0 | 41.7 | 83.3
  Baseline: Normal, Post-Baseline: Mild+ | 0 | 16.7 | 33.3 | 8.3
  Baseline: Normal, Post-Baseline: Moderate+ | 8.3 | 0 | 0 | 0
  Baseline: Normal, Post-Baseline: Mild- | 8.3 | 8.3 | 25.0 | 8.3

12. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Hemoglobin)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 75.0 | 83.3 | 83.3 | 75.0
  Baseline: Normal, Post-Baseline: Mild | 16.7 | 8.3 | 16.7 | 25.0
  Baseline: Normal, Post-Baseline: Moderate | 8.3 | 8.3 | 0 | 0

13. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (White Blood Cell [WBC])
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 91.7 | 83.3 | 66.7 | 83.3
  Baseline: Normal, Post-Baseline: Mild+ | 8.3 | 16.7 | 25.0 | 8.3
  Baseline: Normal, Post-Baseline: Moderate+ | 0 | 0 | 8.3 | 0
  Baseline: Normal, Post-Baseline: Mild- | 0 | 0 | 0 | 8.3

14. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Lymphocytes)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 91.7 | 100.0
  Baseline: Normal, Post-Baseline: Moderate | 0 | 0 | 8.3 | 0

15. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Neutrophils)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 100.0 | 91.7
  Baseline: Normal, Post-Baseline: Severe | 0 | 0 | 0 | 8.3

16. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Eosinophils)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 91.7 | 91.7 | 83.3
  Baseline: Normal, Post-Baseline: Mild | 0 | 8.3 | 8.3 | 16.7

17. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Platelet Count)
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post Baseline: Normal | 100.0 | 100.0 | 100.0 | 100.0
  Baseline:Normal,Post Baseline:Mild/Moderate/Severe | 0.0 | 0.0 | 0.0 | 0.0

18. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Sodium).
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 91.7 | 91.7 | 83.3
  Baseline: Normal, Post-Baseline: Mild+ | 0 | 8.3 | 0 | 0
  Baseline: Normal, Post-Baseline: Moderate+ | 0 | 0 | 0 | 8.3
  Baseline: Normal, Post-Baseline: Severe+ | 0 | 0 | 8.3 | 0
  Baseline: Normal, Post-Baseline: Grade 4 increase | 0 | 0 | 0 | 8.3

19. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Potassium).
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 91.7 | 75.0 | 100.0 | 100.0
  Baseline: Normal, Post-Baseline: Mild+ | 0 | 8.3 | 0 | 0
  Baseline: Normal, Post-Baseline: Grade 4 increase | 8.3 | 16.7 | 0 | 0

20. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Blood Urea Nitrogen [BUN]).
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 100.0 | 100.0
  Baseline:Normal,Post Baseline:Mild/Moderate/Severe | 0.0 | 0.0 | 0.0 | 0.0

21. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Serum Creatinine).
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 100.0 | 100.0
  Baseline:Normal,Post Baseline:Mild/Moderate/Severe | 0.0 | 0.0 | 0.0 | 0.0

22. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Urine Red Blood Cells [RBC]).
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 83.3 | 100.0 | 75.0 | 75.0
  Baseline: Normal, Post-Baseline: Mild | 0 | 0 | 25.0 | 25.0
  Baseline: Normal, Post-Baseline: Moderate | 16.7 | 0 | 0 | 0

23. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Urine Protein).
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 58.3 | 50.0 | 58.3 | 75.0
  Baseline: Normal, Post-Baseline: Mild | 16.7 | 16.7 | 16.7 | 16.7
  Baseline: Normal, Post-Baseline: Moderate | 25.0 | 33.3 | 25.0 | 0
  Baseline: Normal, Post-Baseline: Grade 4 | 0 | 0 | 0 | 8.3

24. Primary Outcome: Percentage of Participants With Change in Severity From Baseline in Laboratory Evaluations (Urine Glucose).
Time Frame: Baseline up to Month 7
Measure: Number; unit: percentage of participants
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
percentage of participants
  Baseline: Normal, Post-Baseline: Normal | 100.0 | 100.0 | 100.0 | 100.0
  Baseline:Normal,Post Baseline:Mild/Moderate/Severe | 0.0 | 0.0 | 0.0 | 0.0

25. Secondary Outcome: Meningococcal Immunoglobulin G (IgG) Geometric Mean Titers (GMT)
Time Frame: Before Dose 1, 1 month after Dose 2, before Dose 3, 1 month after Dose 3
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Number analyzed (Participants) | 12 | 12 | 12 | 12
titers
  Subfamily A: Before Dose 1 (N=12, 12, 12, 12) | 17.3 [6.3 to 47.8] | 16.8 [6.4 to 43.6] | 7.5 [3.1 to 17.8] | 7.9 [3.4 to 18.2]
  Subfamily A: 1 Month After Dose2 (N=10, 12, 11, 9) | 1522.7 [817.5 to 2836.0] | 1933.5 [1036.3 to 3607.6] | 1132.7 [575.0 to 2231.1] | 3.1 [1.7 to 5.5]
  Subfamily A: Before Dose 3 (N=10, 11, 11, 7) | 495.7 [238.0 to 1032.4] | 500.7 [253.6 to 988.7] | 318.6 [147.4 to 688.5] | 3.5 [1.6 to 7.8]
  Subfamily A: 1 Month After Dose 3 (N=8, 10, 9, 7) | 4107.4 [1752.3 to 9627.6] | 4326.9 [2214.5 to 8454.2] | 2664.8 [1410.8 to 5033.4] | 3.8 [2.1 to 6.7]
  Subfamily B: Before Dose 1 (N=12, 12, 12, 12) | 15.6 [6.1 to 40.2] | 7.1 [2.9 to 17.5] | 8.8 [4.0 to 19.5] | 5.1 [2.2 to 12.0]
  Subfamily B: 1 Month After Dose2 (N=10, 12, 11, 9) | 850.5 [547.1 to 1322.2] | 1071.2 [641.4 to 1789.0] | 1300.9 [692.5 to 2443.6] | 2.8 [1.1 to 7.2]
  Subfamily B: Before Dose3 (N=10, 11, 11, 7) | 289.8 [168.0 to 499.8] | 361.4 [192.7 to 677.6] | 370.2 [145.7 to 940.6] | 3.1 [1.1 to 8.8]
  Subfamily B: 1 Month After dose 3 (N=8, 10, 9, 7) | 2081.9 [1098.1 to 3947.1] | 2295.3 [1224.2 to 4303.5] | 3445.0 [1544.9 to 7682.2] | 2.6 [1.0 to 6.8]

ADVERSE EVENTS:
Time Frame: Baseline up to Month 7
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | rLP2086 60mcg | rLP2086 120 mcg | rLP2086 200 mcg | Tdap/Normal Saline (Control)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 11/12 | 11/12 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rLP2086 60mcg (N=12) | rLP2086 120 mcg (N=12) | rLP2086 200 mcg (N=12) | Tdap/Normal Saline (Control) (N=12)
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Induration (General disorders) | 0 | 0 | 1 | 0
Injection site induration (General disorders) | 1 | 1 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 1 | 0 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 6 | 5 | 3
Alanine aminotransferase increased (Investigations) | 2 | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 2 | 6
Blood fibrinogen decreased (Investigations) | 1 | 1 | 2 | 1
Blood fibrinogen increased (Investigations) | 1 | 2 | 6 | 1
Blood potassium increased (Investigations) | 1 | 3 | 0 | 0
Blood sodium increased (Investigations) | 0 | 1 | 1 | 2
Eosinophil count increased (Investigations) | 0 | 1 | 1 | 2
Fibrin D dimer increased (Investigations) | 1 | 3 | 4 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 3 | 2 | 2 | 3
Haemoglobin decreased (Investigations) | 3 | 2 | 2 | 3
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 1 | 0 | 0 | 0
Mean cell haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 1 | 2 | 2 | 2
Platelet count increased (Investigations) | 0 | 1 | 0 | 0
Protein urine (Investigations) | 5 | 6 | 5 | 3
Prothrombin time prolonged (Investigations) | 0 | 0 | 2 | 0
Red blood cell count decreased (Investigations) | 1 | 2 | 1 | 3
Red blood cells urine (Investigations) | 2 | 0 | 2 | 2
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 1
Red cell distribution width increased (Investigations) | 1 | 2 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 1 | 2 | 4 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.